CLINICAL TRIAL: NCT06499883
Title: Agile Development of Innovative, Interactive Hazard Recognition and Mitigation Tools/Learning E-platforms for Workers Involved in Disaster Rescue and Recovery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Principal Investigator, William B Perkison, Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HSC-SPH-23-0741; R44ES030580 (NIH)
Record Dates: First submitted 2023-05-08; First posted 2024-07-15 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Work-related Illness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pocket Ark (Experimental)
  Interventions: Behavioral: Pocket Ark

INTERVENTIONS:
Behavioral: Pocket Ark — Pocket Ark (PA) is a mobile e-learning and assessment platform for use by flood remediation workers in the field. The purpose of this mobile application is to provide workers with real-time data to assist with making safe decisions during the planning phase in the flooded zone and provide a communications platform to improve logistics between operational bases and workers during and after the deployment to the flooded zone. Pocket Ark incorporates an action planner, scenario-based PPE training content, assessments (both knowledge and health-risk), personal security protection, and resource location features for workers involved in disaster rescue and recovery. Individual construction worker's readiness to be safely deployed to flooded and post-flood environments will be assessed.

SUMMARY:
The goal of this study is to assess Pocket Ark (PA), which is a mobile e-learning and assessment platform for use by flood remediation workers in the field. The purpose of the mobile application is to provide workers with real-time data to assist with making safe decisions during the planning phase in the flooded zone and provide a communications platform to improve logistics between operational bases and workers during and after the deployment to the flooded zone. Pocket Ark incorporates an action planner, scenario-based PPE training content, assessments (both knowledge and health-risk), personal security protection, and resource location features for workers involved in disaster rescue and recovery. Individual construction worker's readiness to be safely deployed to flooded and post-flood environments will be assessed.

DETAILED DESCRIPTION:
Enrolled participants will be asked to complete: 1) basic demographic and occupational health information; 2) a simulated wage contract with an employer; 3) a pre-behavioral capability test; and 4) a post flood disaster scenario, which is based on an actual flooding event that has occurred. Participants will be asked questions regarding their response to different challenges he/she might encounter in a post flood construction event and then the correct answer will be provided for learning. Information will be largely graphical, and workers can take the module over the course of several days. Educational material will be based on the Federal Emergency Management Agency (FEMA) Emergency Management Institute and the Center for Construction Research and Training disaster preparedness programs.

Finally, participants will complete: 5) a post behavioral capability test and 6) a brief medical questionnaire of the participant's medical history. Based on the results of the educational testing and the completed medical response, a Readiness Index will be calculated for the participant and relayed to both the participant and the worker advocacy organization. This readiness index will be derived from achieving a passing score of 70% of behavioral capability on the educational and scenario modules, successful completion of the health screening questionnaire, and successful completion of a wage contract.

A brief acceptability assessment and exit interview survey will be completed by participants, and it will assess the program's usefulness, evaluate for technical glitches encountered, request suggestions for future implementation, and derive ratings on PA perceived impact.

Additionally, a worker advocacy staff member who normally conducts disaster preparedness training and a member of the worker advocacy program upper management will be asked to go through the training and answer questions regarding program usability from their perspective.

ELIGIBILITY:
Inclusion Criteria:

* Reconstruction workers
* Affiliated members of the worker advocacy organization
* Professional experience working in the construction industry
* Have a 3- year or newer version cell phone capable of accessing the internet
* Has not completed a Resilience Force training in the last 2 years

Exclusion Criteria:

* inability to complete requested activities
* lack of cell phone connectivity

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2024-07-11 (Estimated); Primary Completion 2024-07-12 (Estimated); Study Completion 2024-07-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants who have increased behavioral capability as assessed by a survey | baseline, after completion of Pocket Ark education (within 2 hours of baseline)
  A survey will be used to assess the worker's procedural knowledge on the steps and skills to negotiate a contract and meet criteria for operational readiness for post-flood clean-up.

SECONDARY OUTCOMES:
Usability of the Pocket Ark mobile application as assessed by the Technology Acceptance Model (TAM) | after completion of Pocket Ark education (within 2 hours of baseline)
  Total score on the Technology Acceptance Model (TAM) ranges from 5 to 25, with a lower the score indicating greater usability.
Usability of the Pocket Ark mobile application as assessed by the System Usability Scale (SUS) | after completion of Pocket Ark education (within 2 hours of baseline)
  Total score on the System Usability Scale (SUS) ranges from 0 to 100, with a higher score indicating greater usability.

CONTACTS AND LOCATIONS:
Overall Officials: William B Perkison, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No